CLINICAL TRIAL: NCT01495650
Title: A Randomized Controlled Trial to Evaluate the Effect of a Tailored Program of Physical Activity and Nutritional Counseling on Fatigue Reduction in Breast Cancer Patients Receiving Adjuvant Treatment.
Brief Title: Effect of a Tailored Program of Physical Activity and Nutritional Counseling on Fatigue Reduction in Breast Cancer Patients Receiving an Adjuvant Treatment
Acronym: APAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APAD; 2010-A00906-33 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2011-12-15; First posted 2011-12-20 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer
Keywords: Comprehensive Adjuvant Care; Cancer-related fatigue; Therapeutic patient education; Physical Activity; Nutritional counselling; Rehabilitation
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention arm (Experimental)
  Interventions: Behavioral: Tailored program of PA and nutritional counseling
- Control arm (No Intervention): Routine practice

INTERVENTIONS:
Behavioral: Tailored program of PA and nutritional counseling — Patients receive tailored program of physical exercises and nutritional counseling during the course of adjuvant treatments (CT followed by RT, 27 weeks).
  Arms: Intervention arm

SUMMARY:
Cancer-related fatigue is by far the most common symptom affecting cancer patients. Combining regular dietary counseling and tailored physical activity is associated with reduced cancer-related fatigue and can improve quality of life and body weight control. We propose to conduct a randomized controlled trial which purpose is to evaluate the effect of an intervention combining physical exercise and nutritional therapeutic education on cancer-related fatigue. To gain behavioral change towards PA and nutrition habits, interventions will take place within hospitals, on the same days of adjuvant treatments.

DETAILED DESCRIPTION:
Cancer-related fatigue is by far the most common symptom affecting cancer patients. Combining regular dietary counseling and tailored physical activity is associated with reduced cancer-related fatigue and can improve quality of life and body weight control. We propose to conduct a randomized controlled trial which purpose is to evaluate the effect of an intervention combining physical exercise and nutritional therapeutic education on cancer-related fatigue. To gain behavioral change towards PA and nutrition habits, interventions will take place within hospitals, on the same days of adjuvant treatments.

ELIGIBILITY:
Inclusion Criteria:

* Female patient with histologically proven breast cancer
* 18-76 years old
* Patients having undergone curative surgery and eligible to 6 cycles of adjuvant chemotherapy (6 FEC100, or 3FEC100 + taxanes) followed by radiotherapy
* Satisfactory healing of breast and lymph nodes area
* Ability to understand the nature, goal and study methodology
* Consent to cooperate for clinical assessments
* Affiliation to a social security regime or beneficiary of equivalent social protection
* Written informed consent provided before any study specific procedures

Exclusion Criteria:

* HER2 positive or metastatic cancer
* Any other primary tumor
* Contraindication to moderate physical activity
* Contraindication to adjuvant chemotherapy or radiotherapy
* Pregnancy or breast feeding
* Inability to attend or comply with interventions or follow-up scheduling, disability or difficulty preventing a proper understanding of trial

Ages: 18 Years to 76 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2010-12; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Subjective fatigue | At 18 months
  Subjective fatigue is measured using the Multidimensional Fatigue Inventory (MFI-20) questionnaire

SECONDARY OUTCOMES:
Quality of life | At 18 months
  Quality of life is measured by the EORTC QLC-C30 questionnaire
Anxiety/depressive symptoms | At 18 months
  Anxiety/depressive symptoms is measured by the HADS questionnaire
Physical activity level | At 18 months
  Physical activity level is measured by the GPAQ questionnaire
Muscular fatigue | At 18 months
  Muscular fatigue is measured by Myotest
Attention fatigue | At 18 months
  Attention fatigue is measured usingt the TAP 2.2 software
Body Mass Index | At 18 months
  Body Mass Index is calculated using bodyweight and length measurements
Body composition | At 18 months
  Body composition (fat mass/fat-free mass ratio) is assessed by dual-energy X-ray absorptiometry (DEXA)

CONTACTS AND LOCATIONS:
Locations (1):
- CRLC Val d'Aurelle-Paul Lamarque, Montpellier, France

REFERENCES:
- [Derived] Touraine C, Jacot W, Gourgou S, Carayol M, Senesse P, Ninot G, Mollevi C. Impact of adapted physical activity and diet counselling on health-related quality of life in women undergoing adjuvant breast cancer therapy. Sci Rep. 2025 Mar 10;15(1):8215. doi: 10.1038/s41598-025-91569-w. PMID 40064980
- [Derived] Carayol M, Ninot G, Senesse P, Bleuse JP, Gourgou S, Sancho-Garnier H, Sari C, Romieu I, Romieu G, Jacot W. Short- and long-term impact of adapted physical activity and diet counseling during adjuvant breast cancer therapy: the "APAD1" randomized controlled trial. BMC Cancer. 2019 Jul 25;19(1):737. doi: 10.1186/s12885-019-5896-6. PMID 31345179